CLINICAL TRIAL: NCT07184008
Title: Echocardiographic and Electrocardiographic Findings in Pediatric Patients With Neurological Findings.
Brief Title: Echo and ECG Findings in Neuropediatrics
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Youssef Qestandy Youssef, Assiut University, Assiut University
Other Study IDs: Ecg & Echo in neuropediatrics
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Migraine Seizures Encephalopathy; Arrythmia Congenital Heart Disease Cardiomyopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the echo-electrocardiographic findings in patients with neurological affection to identify potential cardiac involvement, and explore correlation between cardiac and neurological abnormalities.Objectives are To assess echocardiographic findings in patients with neurological affection , to analyze ECG patterns in the same patient group and to explore clinical significance of detected cardiac findings in the management of neurological patients.

DETAILED DESCRIPTION:
Neurological disorders in pediatric patients represent a significant cause of morbidity and mortality worldwide. These disorders may have multifactorial etiologies , including congenital , infectious , metabolic , inflammatory , and vascular causes , with clinical presentations ranging from seizures to motor deficits and altered consciousness.

The interplay between neurological conditions and cardiovascular involvement has gained increasing attention in recent years. Cardiac manifestations may occur secondary to neurological diseases due to autonomic dysregulation , systemic inflammation , or direct neuro cardiac interaction , potentially affecting patient outcomes.

Several studies have demonstrated that pediatric patients with neurological diseases, such as epilepsy, cerebral palsy, and acute encephalitis, may exhibit significant echocardiographic and electrocardiographic changes. These changes may be transient or persistent, and recognizing them early is crucial for comprehensive patient management.

Moreover, neurological complications may also arise as a consequence of primary cardiac disease. Conditions such as congenital heart disease, infective endocarditis, or shunt lesions can predispose to embolic stroke, brain abscess, or hypoxic-ischemic injury, representing critical intersections between heart and brain.

Electrocardiographic abnormalities are frequently observed in children with congenital and acquired heart disease, and some of these changes are associated with neurological complications. For instance, prolonged QT interval or QT dispersion has been linked to an increased risk of arrhythmia-related cerebral hypoperfusion and syncope, which in turn can precipitate transient ischemic attacks or seizures.

Atrial fibrillation, although less common in children, may also occur in certain congenital heart conditions and cardiomyopathies. It is a well-recognized source of cardioembolic stroke, as thrombi formed in the atria can dislodge and travel to the cerebral circulation. Early detection of such arrhythmias by ECG is essential to prevent neurological sequelae.

Understanding the cardiac profile of patients with neurological affection may therefore help in early detection, appropriate intervention, and reduction of long-term complications.

ELIGIBILITY:
Inclusion Criteria:

1. pediatric patients (1 month - 18 years) diagnosed with a neurological disorder (e.g., stroke, epilepsy, demyelinating disorders, neuromuscular diseases and migraine) confirmed by clinical data (history & examination) and/or neuroimaging ( CT & MRI ).
2. Both sexes (Male & Female) were included in the study.
3. Patients willing to participate and provide informed consent

Exclusion Criteria:

1. patients younger than 1 month old.
2. critically unstable patients in whom echocardiography could not be performed safely or was technically in adequate for interpretation.
3. patients refuse to participate in the research.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population will include pediatric patients presenting with neurological manifestations (such as seizures, motor deficits, stroke, or altered consciousness) who are admitted to the Pediatric Neurology and Cardiology Departments, or presenting to the Emergency Room (ER) at Assiut University Hospital. These patients will be further evaluated for underlying cardiac diseases using echocardiography (ECHO) and electrocardiography (ECG). Both male and female patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Detection of cardiac abnormalities in pediatric patients with neurological disorders | Within the first week of hospital admission
  Proportion of patients showing abnormalities in either electrocardiography (arrhythmias, conduction defects, prolonged QTc) or echocardiography (structural heart disease, ventricular dysfunction, pulmonary hypertension, vegetations).

IPD SHARING:
Plan to Share IPD: Undecided